CLINICAL TRIAL: NCT02874430
Title: A Phase II Study of Metformin in Combination With Doxycycline in Patients With Localized Breast, and Uterine, and Cervical Cancer
Brief Title: Metformin Hydrochloride and Doxycycline in Treating Patients With Localized Breast or Uterine Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.317
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Breast Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Uterine Corpus Cancer; Uterine Corpus Carcinosarcoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (metformin hydrochloride, doxycycline) (Experimental): Patients receive metformin hydrochloride orally daily on days 1-3 and twice a day starting on day 4. Patients also receive doxycycline orally every 12 hours starting on day 1. Treatment repeats every 7 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Metformin Hydrochloride; Drug: Doxycycline

INTERVENTIONS:
Drug: Metformin Hydrochloride — Given orally
  Other Names: 1,1-Dimethylbiguanide Hydrochloride; 1115-70-4; 91485; Cidophage; Dimefor; Glifage; Glucoformin; Glucophage; N,N-Dimethylimidodicarbonimidic Diamide Monohydrochloride; Riomet; Siofor
Drug: Doxycycline — Given orally
  Other Names: 17086-28-1; Doxycycline Monohydrate

SUMMARY:
This phase II trial studies how well metformin hydrochloride works together with doxycycline in treating patients with localized breast or uterine cancer. Metformin hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Doxycycline may stop the growth of bacteria by keeping them from making proteins and minimized the toxic side effects of anti-cancer therapy. It is not yet known whether giving metformin hydrochloride together with doxycycline may be a better way in treating patients with localized breast or uterine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if treatment with a combination of metformin and doxycycline can increase the percentage of cells that express Caveolin-1 in the cancer associated fibroblasts of patients with breast, or uterine, and cervical cancers.

SECONDARY OBJECTIVES:

I. To determine the effect of metformin and doxycycline treatment on the percentage of cells that express monocarboxylate transporter (MCT)4 in cancer associated fibroblasts and MCT1 and transporter of outer mitochondrial membrane (TOMM)20 in the cancer cells of breast and uterine cancer patients.

II. To assess safety and tolerability of metformin and doxycycline treatment in subjects with breast and uterine cancer.

III. To determine the relationship of the percentage of stromal cells expressing caveolin (CAV)1 or MCT4 and tumor cells that express MCT1 and TOMM20 at baseline and after treatment with metformin and doxycycline with the percentage of cells expressing estrogen receptor (ER) and progesterone receptor (PR) for breast and uterine samples and human epidermal growth factor (HER)2 in breast cancer samples.

TERTIARY OBJECTIVES:

I. To assess the effect of combined metformin and doxycycline therapy on the metabolic profile of cancer cells and stroma using mass spectroscopy imaging (MSI) on paired samples, comparing metabolite profiles in the pre-metformin and post-metformin tumor sample.

II. To assess, when possible, the impact of a patient's nutritional status, estimated using 3 day dietary recall versus caloric needs as calculated by the Harris-Benedict equation on the baseline and net change in CAV1 III. To assess the effect of combined metformin and doxycycline therapy on oncomiR micro ribonucleic acid (RNA) (miR-21) after intervention.

IV. To assess the effect of combined metformin and doxycycline therapy on adipokines and the insulin-like growth factor (IGF)-1/insulin signaling pathways through assessment of serum triglycerides, IGF-1, IGF-binding protein (BP)3, erythrocyte sedimentation rate (ESR), adiponectin, leptin, IGF-1 receptor (R), exosome evaluation, metabolomics profile, and microRNA expression profile.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Diagnosis of localized breast or uterine cancer that is either biopsy proven or suspected based on history, physical, and or radiographic findings, and who are planned for definitive resection of the tumor without the use of neoadjuvant chemotherapy or radiation therapy at TJUH are eligible to participate.
2. Subjects must be ≥ 18 years of age at time of consent.
3. Subjects must be newly diagnosed or suspected to have breast, uterine (endometrial cancer with histologies including endometrioid, serous, clear cell, and carcinosarcoma) or cervical cancer.
4. Patient must be able to swallow pills.
5. Patients with serum creatinine levels less than 1.5 mg/dL.
6. Women of child bearing potential must have a negative urine or blood pregnancy test within 14 days of study enrollment.
7. Informed Consent: All subjects must be able to comprehend and sign a written informed consent document.
8. ECOG Performance status <1

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Received any prior cancer therapy for the breast or uterine cancer that is being resected, including progesterone therapy for endometrial cancer patients.

   a. Patients may have had prior therapy for other contra-lateral breast cancer.
2. Subjects who are pregnant or breastfeeding or may become pregnant during metformin and doxycycline administration.
3. Subjects on metformin or doxycycline for any reason during the preceding 4 weeks.
4. Diabetic subjects that are managed by taking metformin or insulin.
5. Subjects who have received iodinated contrast dye must wait 12 hours prior to starting Metformin. If a CT scan with contrast is scheduled after screening and consent, the metformin cannot be taken until after the CT with contrast has been completed and they have waited 12 hours.
6. Patients with serum creatinine level greater than 1.5 mg/dL.
7. Patients with history of lactic or any other metabolic acidosis.
8. Patients with history of congestive heart failure stage III or greater.
9. Patients scheduled for definitive cancer surgical resection less than 7 days from beginning of study drug administration or greater than 6 weeks from beginning study drug administration.
10. Patients with history of hepatic dysfunction or hepatic disease and abnormal liver function tests defined as AST, ALT, Alk Phos, and or total bilirubin greater than 2.5 times the upper limit of normal.

    a. Patients who have a history of hepatic dysfunction or hepatic disease and normal liver function tests will be eligible to participate.
11. Patients with a current history (in the past 30 days) of heavy drinking which is defined in accordance with CDC definition as more than 8 drinks per week for women and more than 15 drinks per week for men. A standard drink contains .6 ounces of pure alcohol. Generally, this amount of pure alcohol is found in 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor (e.g., gin, rum, vodka, or whiskey). While on study, patients should limit their alcohol consumption to no more than 8 drinks per week for women and no more than 15 drinks per week for men. Patients who feel they cannot comply with this recommendation are not eligible.
12. Prior allergic reaction to metformin, doxycycline, or any other tetracycline antibiotic in the past.
13. Patient is on medications that are contraindicated with metformin or doxycycline under current FDA recommendations. The following is a list of medications identified as class D (consider therapy modification) when treatment with metformin or doxycycline is considered:

    * Class D:

      * Bismuth Subsalicylate
      * Cimetidine
      * Iodinated contrast agents
      * Somatropin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in the percent of stromal cells expressing Caveolin-1 (CAV1) at an intensity of 1+ or greater assessed by immunohistochemistry | Baseline to week 6
  Within-patient change in immunohistochemistry scores will be analyzed using the Wilcoxon signed-rank test.

SECONDARY OUTCOMES:
Incidence of adverse events evaluated using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | At 30 days after last dose of metformin and doxycycline
Change in the percent of stromal cells expressing express Monocarboxylate Transporter 4 (MCT4) in the cancer cells | Baseline up to week 5
  Analysis will be performed separately in breast and uterine cancer patients. Evaluated using Aperio analyses of expression intensity with previously validated algorithms. Analysis will be performed using the Wilcoxon signed-rank test.
Change in the percent of tumor cells that express Monocarboxylate Transporter 1 (MCT1) and Transporter of Outer Mitochondrial Membrane 20 (TOMM20) in the cancer cells | Baseline up to week 5
  Analysis will be performed separately in breast and uterine cancer patients. Evaluated using Aperio analyses of expression intensity with previously validated algorithms. Analysis will be performed using the Wilcoxon signed-rank test.
Percentage of stromal cells expressing Caveolin-1 (CAV1) or Monocarboxylate Transporter 4 (MCT4) | Baseline up to week 5
  Assessed in relation to the percentage of cells expressing Estrogen Receptor (ER) and Progesterone Receptor (PR) for breast and uterine samples and Human Epidermal Growth Factor Receptor 2 (HER2) in breast cancer samples.
Percentage of tumor cells that express Monocarboxylate Transporter 1 (MCT1) and Transporter of Outer Mitochondrial Membrane 20 (TOMM20) | Baseline up to week 5
  Assessed in relation to the percentage of cells expressing Estrogen Receptor (ER) and Progesterone Receptor (PR) for breast and uterine samples and Human Epidermal Growth Factor Receptor 2 (HER2) in breast cancer samples.
Progress-free survival | Up to 12 months post last dose of metformin and doxycycline
  Will be estimated using the Kaplan-Meier method.
Overall survival | Up to 12 months post last dose of metformin and doxycycline
  Will be estimated using the Kaplan-Meier method.
Objective response rate | Up to 12 months post last dose of metformin and doxycycline
  Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/